CLINICAL TRIAL: NCT01497041
Title: A Phase II Clinical Trial of Docetaxel, Oxaliplatin Combination Chemotherapy in Patients With Stage IIIB/IV Non-adenocarcinoma, Non-small Cell Lung Cancer (NSCLC) as Second-line Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean South West Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSWOG 2010-3
Record Dates: First submitted 2011-12-14; First posted 2011-12-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous; Carcinoma, Large Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Carcinoma, Large Cell | interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Docetaxel — Docetaxel (diluted in 250 ml of 5% dextrose solution, over 60 minutes) 35 mg/m2 IV (D1, D8) every 3 weeks
Drug: Oxaliplatin — Oxaliplatin (diluted in 500 ml of 5% dextrose solution, over 120 minutes) 60 mg/m2 IV D1 every 3 weeks

SUMMARY:
1. Goals

   The primary goal of this phase II trial is to:

   evaluate the response rate of combination chemotherapy with docetaxel and oxaliplatin in patients with stage IIIB/IV non-adenocarcinoma, non-small cell lung cancer (NSCLC) as second-line treatment

   Secondary goals are to:

   evaluate the treatment-related toxicities of this combination, investigate progression-free survival (PFS) and overall survival (OS) in this population
2. Design The proposed clinical trial is an open label, non-comparative, multicenter phase II trial according to the two stage testing design by Simon two-stage testing procedure

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed as non-adenocarcinoma, non-small cell carcinoma of lung histologically or cytologically
2. Patients must be ≥ 18 years old of age
3. ECOG performance status ≤ 1
4. Estimated life expectancy of more than 3 months
5. Treatment with only one prior chemotherapy
6. At least one lesion that can be measured by imaging (CT/MRI) according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
7. Adequate bone marrow function (absolute neutrophil count [ANC] ≥ 1,500/µL, hemoglobin ≥ 9.0 g/dL [correction by transfusion is acceptable], and platelets ≥ 100,000/µL)
8. Adequate kidney function (serum creatinine < 1.5 x upper limit of normal [ULN])
9. Adequate liver function (serum total bilirubin < 1.5xULN; serum transaminases levels < 2.5xUNL)
10. Provision of fully informed consent prior to any study specific procedures

Exclusion Criteria:

1. Pregnant or breastfeeding women and women of childbearing potential not employing adequate contraception
2. Patients who received prior chemotherapy including paclitaxel or docetaxel
3. Patients with second primary cancer (except, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥5 years)
4. Patients with defect of central nervous system (CNS) or any psychiatric disorders and CNS metastases
5. Other serious illness or medical conditions A. Clinically significant cardiac disease (uncontrolled congestive heart disease despite treatment [NYHA class III or IV], symptomatic coronary artery disease, unstable angina or myocardial infarction, conduction abnormality like grade 2 AV block, serious arrhythmia needed for medication, uncontrolled hypertension) within 6 months prior to study entry B. Liver cirrhosis (≥ Child-Pugh class B) C. History of significant neurologic or psychiatric disorders including dementia or seizures D. Active uncontrolled infection E. Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
6. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2years
  Assessment of response will be assessed according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Overall survival | 2years
  Overall survival will be calculated by Kaplan-Meier method
Progression free survival | 2 years
  Progression free survival will be calculated by Kaplan-Meier method
Number of Participants with Adverse Events | 2 years
  Assessment of toxicity will be assessed according to CTCAE version 4.0
Quality of life | 2 years
  Quality of life will be assessed according to EORTC QLQ-C30, LC13

CONTACTS AND LOCATIONS:
Overall Officials: Sang Byung Bae, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (5):
- South Korea (5):
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea Daejeon ST. Mary's Hospital, Daejeon
  - Chonbuk National University Hospital, Jeonju